CLINICAL TRIAL: NCT05953350
Title: A Phase Ib/II Study Confirmed Inhibition of Autophagy Synergizes Anti-tumor Effect of High Dose CDK4/6i with Manageable Safety in HR+HER2-breast Cancer Patients
Brief Title: A Phase Ib/II Study Confirmed Inhibition of Autophagy Synergizes Anti-tumor Effect of High Dose CDK4/6i
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Gong, Prof., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SKSKY-2023-488-01
Record Dates: First submitted 2023-06-12; First posted 2023-07-20 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Inhibition of Autophagy Synergizes Anti-tumor Effect
Keywords: inhibition of autophagy; CDK4/6i; hydroxychloroquine; HR+HER2-breast cancer
MeSH Terms: interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase Ib clinical trial (Experimental): 600mg bid dose of hydroxychloroquine group combined with three predefined dose groups of palbociclib: 100mg QD, 150mg QD, and 200mg QD, separately.
  Interventions: Drug: 600mg bid dose of hydroxychloroquine combined with three predefined dose groups of palbociclib
- Phase II clinical trial (Experimental): After MTD was determined, RP2D dose was selected for phase II clinical trial.
  Interventions: Drug: RP2D dose of 600mg bid of hydroxychloroquine combined with palbociclib was selected for phase II clinical trial.

INTERVENTIONS:
Drug: 600mg bid dose of hydroxychloroquine combined with three predefined dose groups of palbociclib — hydroxychloroquine group of 600mg bid combined with three predefined dose groups of palbociclib: 100mg QD, 150mg QD, and 200mg QD, separately.
  Arms: Phase Ib clinical trial
Drug: RP2D dose of 600mg bid of hydroxychloroquine combined with palbociclib was selected for phase II clinical trial. — After the exploration of 600mg bid dose of hydroxychloroquine combined with palbociclib, and the maximal tolerated dose (MTD) was determined, then RP2D dose of 600mg bid dose of hydroxychloroquine combined with palbociclib was selected for phase II clinical trial.
  Arms: Phase II clinical trial

SUMMARY:
In order to explore the safety and antitumor efficacy of different doses of CDK4/6 inhibitor Palbociclib in combination with the autophagy inhibitor hydroxychloroquine (HCQ) , a phase Ib/II study was conducted.

This study will adopt a 3+3 design and include three predefined dose groups of palbociclib: 100mg QD, 150mg QD, and 200mg QD. Initially, 600mg bid dose of hydroxychloroquine group will be administered in combination. The trial will use the first cycle (28 days) as the observation period for tolerability, observing and evaluating the occurrence of DLTs after medication and determining the maximum tolerated dose/maximum administered dose (MTD/MAD) and recommended phase 2 dose (RP2D) of the combination therapy.

This study improves the efficacy of CDK4/6 inhibitors in the treatment of solid tumors by reversing DTP status through the use of HCQ.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with advanced solid tumors (including breast cancer, undifferentiated liposarcoma, etc.) confirmed by histology and/or cytology, who have failed CDK4/6 inhibitor treatment or have experienced failure of neoadjuvant or adjuvant CDK4/6 inhibitor therapy for 12 months.
2. At least one measurable target lesion according to RECIST 1.1.
3. Age 18 years or older, any gender.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Expected survival of at least 3 months.
6. Within one week before enrollment, baseline blood tests should be essentially normal (no blood transfusions or hematopoietic growth factor treatment within 14 days): absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; hemoglobin ≥ 9 g/dL; platelet count (PLT) ≥ 75 × 10^9/L.
7. Within one week before enrollment, baseline liver and kidney function tests should be essentially normal (normal values determined by each study center's laboratory): total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); serum glutamic-pyruvic transaminase (SGPT/ALT) ≤ 3 × ULN (≤ 5 × ULN for patients with liver metastases or liver cancer); serum glutamic-oxaloacetic transaminase (SGOT/AST) ≤ 3 × ULN (≤ 5 × ULN for patients with liver metastases); serum creatinine ≤ 1.5 × ULN or creatinine clearance (Ccr) ≥ 50 ml/min.
8. Fertile patients (both males and females) must agree to use a reliable contraceptive method concurrently with their partners during the trial and for at least 3 months after the last dose of medication (hormonal or barrier methods, or abstinence). Pre-menopausal female patients must have a negative pregnancy test in blood or urine before enrollment.
9. Pre-menopausal women should provide blood and urine samples to confirm a negative pregnancy status and commit to using contraception during the study period and for 6 months after the study. Male participants are required to commit to using contraception with their partners or female partners during the study period and for 6 months after the study.

Exclusion Criteria:

1. Patients who have undergone major visceral surgery (excluding needle biopsies) or significant trauma within 4 weeks prior to the first administration of the study drug.
2. Prior treatment with radiotherapy and two or more CDK4/6 inhibitors for advanced or metastatic disease.
3. Failure to recover from adverse reactions of previous anti-tumor therapy to CTCAE 5.0 grade ≤ 1 (except for acceptable toxicities without safety risks, such as hair loss, and manageable immune-related adverse reactions). Additionally, symptomatic peripheral neuropathy of CTCAE 5.0 grade ≥ 2 resulting from the previous treatment regimen.
4. Clinical symptoms of central nervous system metastases or leptomeningeal metastases, or other evidence indicating uncontrolled central nervous system metastases or leptomeningeal metastases deemed unsuitable for enrollment by the investigator.
5. Pregnancy (positive pregnancy test) or lactation.
6. Active infection requiring systemic antimicrobial therapy that is not under control at present (except for asymptomatic urinary tract infections). History of immune deficiency, including positive HIV antibody testing. History of active hepatitis B (except for controlled cases with antiviral therapy) and positive hepatitis C antibody.
7. History of severe cardiovascular or cerebrovascular diseases, including but not limited to clinically significant cardiac rhythm or conduction abnormalities requiring clinical intervention, ventricular arrhythmias, second- or third-degree atrioventricular block; average QTcF > 470 ms based on three consecutive 12-lead electrocardiograms at rest; acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular events within 6 months before the first dose; uncontrolled hypertension.
8. Patients with psychiatric disorders or poor compliance.
9. Patients unsuitable for hydroxychloroquine use due to the presence of retinal vascular disease.
10. Other systemic medical history or conditions deemed inappropriate for participation in the trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The safety dose of the combination of hydroxychloroquine and CDK4/6 inhibitors in patients | 12 months
  The study aims to evaluate the safety dose of the combination of hydroxychloroquine and CDK4/6 inhibitors in patients with solid tumors. The safety dose was according to "3+3" dose escalation principle.
  In this study, Dose-limiting toxicity (DLT) was defined as drug-related adverse reactions (according to the NCI CTC 5.0 grading criteria) after treatment: ≥ Grade II liver and kidney injury, grade III other non-hematological toxicity, and grade IV hematological toxicity.
the recommended phase II dose | 12 months
  The study aims to evaluate the recommended phase II dose of the combination of hydroxychloroquine and CDK4/6 inhibitors in patients with solid tumors.

SECONDARY OUTCOMES:
Objective response rate（ORR） | 12 months
  This study investigates the preliminary efficacy of the combination of hydroxychloroquine and CDK4/6 inhibitors in the treatment of solid tumors.
Progression-free survival (PFS) | 12 months
  This study investigates the preliminary efficacy of the combination of hydroxychloroquine and CDK4/6 inhibitors in the treatment of solid tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong C, Lin Q, Qin T, Zeng Y, Xu F, Yang Y, Yin D, Duan Z, Chen CL, Wing-Cheong Chow L, Liu Q, Hamai A, Mehrpour M, Lin Q, Li J, Song E. Targeting autophagy plus high-dose CDK4/6 inhibitors in advanced HR+HER2- breast cancer: A phase 1b/2 trial. Med. 2025 May 9;6(5):100559. doi: 10.1016/j.medj.2024.11.012. Epub 2024 Dec 27. PMID 39731909